CLINICAL TRIAL: NCT03553498
Title: Randomized Clinical Trial of IV Acetaminophen as an Adjuvant Analgesic to IV Hydromorphone for Treatment of Acute Severe Pain in Non-Elderly Emergency Department Patients
Brief Title: IV Acetaminophen as Adjuvant Analgesic to Hydromorphone - Emergency Department Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Polly Bijur, Professor of Emergency Medicine, Epidemiology and Population Health, and of Pediatrics, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-8886
Record Dates: First submitted 2018-05-10; First posted 2018-06-12 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Acute Pain
Keywords: pain; opioid analgesics; Emergency Department; randomized controlled trial; acetaminophen; hydromorphone
MeSH Terms: conditions — Acute Pain; Pain; Emergencies | interventions — Acetaminophen; Saline Solution; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist working in an area inaccessible to ED staff will ensure blinding by creating identical vials containing either 1000 mg acetaminophen in 100 ml normal saline or 100 ml normal saline placebo and numbering them sequentially for use in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV hydromorphone and IV acetaminophen (Experimental): 1000 mg IV acetaminophen administered over 5-10 minutes
  1 mg hydromorphone administered over 5-10 minutes
  Interventions: Drug: IV acetaminophen; Drug: hydromorphone
- IV hydromorphone and placebo (Placebo Comparator): 100 ml IV normal saline administered over 5-10 minutes
  1 mg hydromorphone administered over 5-10 minutes
  Interventions: Drug: IV placebo; Drug: hydromorphone

INTERVENTIONS:
Drug: IV acetaminophen — acetaminophen given intravenously
  Other Names: Ofirmev
  Arms: IV hydromorphone and IV acetaminophen
Drug: IV placebo — given intravenously
  Other Names: normal saline
  Arms: IV hydromorphone and placebo
Drug: hydromorphone — hydromorphone given intravenously
  Other Names: Dilaudid

SUMMARY:
The goal of this randomized clinical trial is to compare the analgesic efficacy and side effect profile of IV acetaminophen as an analgesic adjunctive medication to IV hydromorphone for the treatment of acute pain experienced by patients in the Emergency Department (ED).

DETAILED DESCRIPTION:
Multimodal treatment of pain is a commonly used strategy to control pain by combining analgesics with different and complementary mechanisms of action. Oral acetaminophen combined with opioids is a mainstay of treatment of mild to moderate pain, while the use of IV opioids is the standard for treatment of severe pain in the Emergency Department. An IV formulation of acetaminophen is widely used in Europe and has recently been approved in the US. It has been studied for treatment of acute post-operative pain and renal colic.

This randomized trial was designed to assess the effectiveness of the combination of IV acetaminophen and IV hydromorphone as a strategy to provide more effective treatment of acute severe pain in the Emergency Department with the possibility of reducing opioid consumption. All patients received 1 mg of IV hydromorphone. They were then randomized to receive either 1 g of IV acetaminophen or 100 mL of normal saline placebo. Measures of pain, vital signs, and presence of side effects were obtained immediately before IV hydromorphone was administered. Following receipt of the acetaminophen or placebo these same variables were measured at 15 minute intervals for the next 120 minutes. Additional analgesics were administered if patients requested them. Subsequent care of the patients was at the discretion of the treating attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Pain with onset within 7 days of the ED visit
* ED attending physician's judgment that the patient's pain warrants IV opioids.
* ED attending physician's judgment that the patient has capacity to provide informed consent.
* ED attending physician's judgement that patient is not a chronic user of opioids or acetaminophen
* Patients must be able to understand English or Spanish.

Exclusion Criteria:

* Use of opioids or tramadol within past 24 hours.
* Use of acetaminophen or non-steroidal anti-inflammatory medication within the previous 8 hours.
* Prior adverse reaction to opioids or acetaminophen.
* Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months; examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies.
* Medical condition that might affect metabolism or opioid analgesics or acetaminophen such as hepatitis, renal insufficiency or failure, hypo- or hyper-thyroidism, Addison's or Cushing's disease
* Pregnant or breastfeeding
* Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician or nurse
* Not at risk of suicide assessed by triage nurse
* Systolic blood pressure <100 mmHg
* Heart Rate < 60/min
* Oxygen saturation < 95% on room air:
* Use of monoamine oxidase (MAO) inhibitors in past 30 days
* Use of transdermal pain patches
* Taking any medication that might interact with one of the study medications, such as a selective serotonin reuptake inhibitor (SSRI) or tricyclic anti-depressants, antipsychotics, anti-malarial medications (quinidine or halofantrine), amiodarone or dronedarone, diphenhydramine, celecoxib, ranitidine, cimetidine, ritonavir, terbinafine or St. John's Wort.
* Patients who have been previously enrolled in this same study

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Polly Bijur, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Hydromorphone and IV Acetaminophen: 1000 mg IV acetaminophen administered over 5-10 minutes
  IV acetaminophen: acetaminophen given intravenously
  1 mg hydromorphone: hydromorphone given intravenously
- IV Hydromorphone and Placebo: 100 ml IV normal saline administered over 5-10 minutes
  IV placebo: given intravenously
  1 mg hydromorphone: hydromorphone given intravenously
Period: Overall Study
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo
Started | 81 | 81
Completed | 80 | 79
Not Completed | 1 | 2
Not completed — Missing primary outcome | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.0) | 43.1 (13.5) | 43.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 28 | 31 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Hispanic/Latino | 54 | 53 | 107
  Race/ethnicity: African-American | 22 | 17 | 39
  Race/ethnicity: White | 2 | 5 | 7
  Race/ethnicity: Other | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 80 | 79 | 159
Location of Pain [Count of Participants; unit: Participants]
  Abdomen/flank | 70 | 67 | 137
  Other | 10 | 12 | 22
Pain Intensity on Numerical Rating Scale [Count of Participants; unit: Participants] — Patient report of pain intensity on Numerical Rating Scale on which 0 = no pain, 10 is worst possible pain
  Participants
    6-7 | 7 | 8 | 15
    8 | 12 | 19 | 31
    9 | 11 | 9 | 20
    10 | 50 | 43 | 93
Nauseated or vomited in Emergency Department before treatment [Count of Participants; unit: Participants]
  Yes - nauseated or vomited | 57 | 52 | 109
  No - not nauseated, did not vomit | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Rating Scale of Pain (NRS) Before Treatment to 60 Minutes After Treatment
Description: The between group difference in change in NRS pain scores from before administration of study medications to 60 minutes post administration of study medications. The NRS is a previously validated and reproducible measure of pain intensity ranging from 0 = no pain, to 10 = worst possible pain. Higher values indicate more pain relief from before treatment to 60 minutes after treatment
Time Frame: Before treatment to 60 minutes after treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo
Number analyzed (Participants) | 80 | 79
units on a scale | 6.2 [5.6 to 6.8] | 5.4 [4.7 to 6.1]
Statistical Analysis 1: Comparison: IV Hydromorphone and IV Acetaminophen vs IV Hydromorphone and Placebo; Test type: Superiority; p = 0.08, t-test, 2 sided

2. Secondary Outcome: Percentage of Patients Who Received Additional Pain Medication Within 60 Minutes of Administration of Study Medication
Description: Difference in percentage of patients who received additional pain medication within 60 minutes of administration of study medication in the two arms of the study
Time Frame: Baseline to 60 minutes post-baseline
Population: All patients in the study
Measure: Count of Participants; unit: Participants
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo
Number analyzed (Participants) | 80 | 79
Participants | 2 | 2
Statistical Analysis 1: Comparison: IV Hydromorphone and IV Acetaminophen vs IV Hydromorphone and Placebo; Test type: Superiority; p = 0.989, Chi-squared

3. Secondary Outcome: Percentage of Patients Who Received Additional Pain Medication Between 61 and 120 Minutes After Administration of Study Medications
Description: Difference in percentage of patients who received additional pain medication between 61 and 120 minutes after administration of study medication by study group
Time Frame: 61 to 120 minutes post-baseline
Population: All patients in study
Measure: Count of Participants; unit: Participants
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo
Number analyzed (Participants) | 80 | 79
Participants | 2 | 4
Statistical Analysis 1: Comparison: IV Hydromorphone and IV Acetaminophen vs IV Hydromorphone and Placebo; Test type: Superiority; p = 0.414, Chi-squared

4. Secondary Outcome: Percentage of Patients Who Want Additional Analgesics
Description: Number of patients who answer "yes" to question: "Do you want more pain medication" divided by number of patients
Time Frame: Immediately after administration of study medication to 120 minutes after administration of study medication
Population: Patients who were still in Emergency Department 120 minutes after medication was administered
Measure: Count of Participants; unit: Participants
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo
Number analyzed (Participants) | 78 | 77
Participants | 21 | 29
Statistical Analysis 1: Comparison: IV Hydromorphone and IV Acetaminophen vs IV Hydromorphone and Placebo; Test type: Superiority; p = 0.153, Chi-squared

ADVERSE EVENTS:
Time Frame: During the entire study - within 2 hours after administration of study medication
Arm/Group | IV Hydromorphone and IV Acetaminophen | IV Hydromorphone and Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/79
Other Adverse Events (participants affected / at risk) | 21/80 | 22/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Hydromorphone and IV Acetaminophen (N=80) | IV Hydromorphone and Placebo (N=79)
Oxygen Desaturation (General disorders) | 3 (3) | 1 (1) — Oxygen saturation less than 95%
Hypotension (General disorders) | 1 (1) | 1 (1) — Systolic blood pressure less than 100 mm Hg
Bradycardia (General disorders) | 0 (0) | 1 (1) — Heart rate less than 50 beats per minute
Nausea and/or Vomiting (General disorders) | 6 (6) | 8 (8)
Pruritis (General disorders) | 11 (11) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT03553498/Prot_SAP_000.pdf